CLINICAL TRIAL: NCT02672306
Title: Clinical Study on the Safety and Efficacy of Umbilical Cord Mesenchymal Stem Cell Injection in the Treatment of Mild and Moderate Alzheimer's Disease
Brief Title: Safety and Exploratory Efficacy Study of UCMSCs in Patients With Alzheimer's Disease
Acronym: SEESUPAD
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South China Research Center for Stem Cell and Regenerative Medicine (Other)
Collaborators: Guangzhou General Hospital of Guangzhou Military Command of PLA (Unknown); Third Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UCMSC-1; NCT02513706 (obsolete NCT alias)
Record Dates: First submitted 2016-01-24; First posted 2016-02-03 (Estimated); Last update posted 2018-04-26 (Actual); Status verified 2018-02

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- UCMSCs (Experimental): Subjects with Alzheimer's Disease Intervention: UCMSCs
  Interventions: Biological: UCMSCs
- Placebo (Placebo Comparator): Subjects with Alzheimer's Disease Intervention: Placebo (normal saline)
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: UCMSCs — Biological: Human UCMSCs 20 million cells per subject (0.5×10^6 UCMSCs per kg) intravenous injection Infusion number: 8 (Once every two weeks)
  Other Names: Human Umbilical Cord Derived Mesenchymal
  Arms: UCMSCs
Biological: Placebo — Subjects with Alzheimer's Disease placebo comparator (normal saline) intravenous injection Infusion number: 8 (Once every two weeks)
  Arms: Placebo

SUMMARY:
The primary purpose of this study is to evaluate the safety and the efficacy of (Human Umbilical Cord-Derived Mesenchymal Stem Cells) UCMSCs for patients with Alzheimer's disease (AD).

DETAILED DESCRIPTION:
Study Type: Interventional Study Design: Treatment, Parallel Assignment, Double Blind (Subject, Outcomes Assessor), Randomized, Safety/ Efficacy Study Official Title: Multicenter, Randomized, Double-blind, Placebo Controlled Trial of UCMSCs in Subjects With Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria:

* Ages 50 to 80, male and female.
* A diagnosis of probable AD and Mixed Dementia according to the criteria of the NINCDS-ADRDA
* Treatment with other cholinesterase inhibitors, such as a stable dose of donnepiazide tablets (5mg/ day or 10mg/ day) or the use of heavy tartaric acid karbalin capsules, is currently being used.
* MMSE score between 10 and 26.
* Voluntarily participating subject who sign the Inform Concent

Exclusion Criteria:

* Caused by other reasons of dementia (vascular dementia, infectious disease of the central nervous system (such as HIV, syphilitic dementia), g - she's disease, Parkinson's disease, Lou gehrig's disease, huntington's disease DLB, traumatic brain dementia, other physical and chemical factors (such as: drug poisoning, alcoholism, carbon monoxide poisoning and other dementia), important body disease (such as hepatic encephalopathy, pulmonary encephalopathy dementia), intracranial placeholder lesions, endocrine system disease, such as thyroid disease, parathyroid disease), and vitamins and other causes of dementia)
* The Hamilton depression scale (HAMD) score > 17, or patients with a history of depression or other psychiatric or psychiatric disorders.
* The Hachinski ischemic index scale (HIS) scored > 4.
* The brief intelligence status examination scale (MMSE) score of 10 patients.
* Liver function (ALT, AST) exceeded the normal range limit of 1.5 times, SCr exceeded normal range upper limit, white blood cell count < 4.0 x 109/L or platelet < 100 x 109/L, hemoglobin < 100g/L.
* Patients with type 1 diabetes, obstructive pulmonary disease (copd) or asthma, vitamin B12 or folate deficiency patients, not control good digestion, liver, kidney, endocrine and cardiovascular system diseases (especially sick sinus syndrome and conduction block), patients with HIV/AIDS, syphilis, active tuberculosis, etc.
* A person with cancer or a history of cancer.
* People with a clinically significant history of stroke, who have had a seizure or a head injury in the past two years, have caused the disorder.
* There is a history of congestive heart failure or a history of myocardial infarction, and a blood disease in two years.
* Drug clinical trials were performed within 3 months of screening.
* Anti-ad agents are being used in addition to the programme requirements.
* The use of stem cell therapy in half a year.
* People with history of alcoholism and substance abuse, allergies, or history of allergies.
* Patients who had been hospitalized for more than 3 months before screening. of allergies.
* The researchers think it is inappropriate to participate in this clinical trial.

Ages: 50 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)Score | 36 weeks from post-administration
  A psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis.

SECONDARY OUTCOMES:
Change in Alzheimer's Disease Assessment Scale - Cognitive Subscale (ADAS-Cog)Score | 10 weeks,18 weeks,24 weeks,48weeks from post-administration
  A psychometric instrument that evaluates memory, attention, reasoning, language, orientation, and praxis.
Change in Mini-Mental State Examination (MMSE) Score | 10 weeks,18 weeks,36 weeks，24 weeks,48weeks from post-administration
  A frequently used screening instrument for Alzheimer's disease drug studies. It evaluates orientation, memory, attention, concentration, naming, repetition, comprehension, and ability to create a sentence and to copy two intersecting polygons.
Change in Clinician's Interview-Based Impression of Change (CIBIC-plus) Score | 10 weeks,18 weeks,24 weeks,36 weeks，48weeks from post-administration
Change in Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory (ADCS-ADL) Score | 10 weeks,18 weeks,24 weeks,36 weeks，48weeks from post-administration
  ADCS-ADL assesses functional performance in subjects with Alzheimer's disease. In a structured interview format, informants are queried as to whether subjects attempted each item in the inventory during the prior 4 weeks and their level of performance. The ADCS-ADL scale discriminates well between normal controls and mild AD patients. It has good test-retest reliability. The ADCS-ADL includes some items from traditional basic ADL scales (e.g., grooming, dressing, walking, bathing, feeding, toileting) as well as items from instrumental activities of daily living scales (e.g., shopping, preparing meals, using household appliances, keeping appointments, reading).
Change in Neuropsychiatric Inventory (NPI) Score | 10 weeks,18 weeks,24 weeks,36 weeks，48weeks from post-administration
  The NPI is a well-validated, reliable, multi-item instrument to assess psychopathology and behavior in AD based on interview with the informant.
Changes in AD Biomarkers | 36 weeks from post-administration
  Plasma beta-amyloid proteins will be collected from blood samples obtained.

OTHER OUTCOMES:
Symptoms Checklist and Adverse Event Assessment | From Day0（administration）to 48 weeks post-administration.
  Adverse events and symptoms checklist are used to monitor signs or symptoms that may or may not be related to study medication, abnormalities detected during physical examination, or clinical significant laboratory abnormalities.

CONTACTS AND LOCATIONS:
Locations (1):
- South China Research Center for Stem Cell and Regenerative Medicine,South China Institute of Biomedicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes